CLINICAL TRIAL: NCT04677192
Title: Effectiveness and Safety Evaluation of Microwave Ablation Combined With Chemotherapy in the Treatment of Pancreatic Cancer Oligohepatic Metastasis: A Prospective, Single-center, Single-arm, Phase II Clinical Study
Brief Title: Microwave Ablation Combined With Chemotherapy in the Treatment of Pancreatic Cancer Oligohepatic Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCLM-A 2020
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Pancreatic Cancer Metastatic to Liver; Oligometastasis
Keywords: Pancreatic Cancer Metastatic to Liver; Oligometastasis; Microwave Ablation; overall survival
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Microwave Ablation Combined with Chemotherapy (Experimental): All patients will receive microwave ablation of oligohepatic metastasis and chemotherapy according to NCCN guidelines,and the efficacy was evaluated every 8 weeks until the disease progressed or the patient could not tolerate it.
  Interventions: Combination Product: Microwave Ablation combination with chemotherapy

INTERVENTIONS:
Combination Product: Microwave Ablation combination with chemotherapy — Microwave Ablation combination with chemotherapy. Maximum tumor diameter ≤ 3cm, single microwave needle, maximum tumor diameter> 3cm, double ablation needle, the ablation range completely covers the lesion ≥ 0.5cm in order to obtain a satisfactory ablation margin. After the operation, contrast ultrasound is performed again to confirm the ablation edge. Enhanced MRI or CT to evaluate the ablation effect 4 weeks after surgery. Selection of chemotherapy regimen refers to the 2020 NCCN Guidelines for Pancreatic Cancer. First-line chemotherapy regimen: gemcitabine combined with albumin-bound paclitaxel or FOLFIRINOX; second-line chemotherapy regimen: If first-line chemotherapy based on gemcitabine, 5-FU-based regimen for second-line, If 5-FU-based regimen for first-line, gemcitabine for second-line.

SUMMARY:
This study is a prospective, single center, single arm, phase II clinical study in patients with liver metastasis after radical resection of pancreatic cancer. The purpose of this study is to evaluate the clinical value of microwave ablation combined with chemotherapy for liver metastasis after radical resection of pancreatic cancer about overall survival, and to determine the feasibility and safety of the scheme.

DETAILED DESCRIPTION:
Microwave ablation, as one of the important treatment methods of liver metastases, has the advantages of radical effect, small trauma and rapid recovery.Microwave ablation combined with chemotherapy aims to improve the quality of life and prolong the survival time.The purpose of this study is to evaluate the clinical value of microwave ablation combined with chemotherapy for liver metastasis after radical resection of pancreatic cancer about overall survival, and to determine the feasibility and safety of the scheme.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75years old, male or female;
* ECOG PS: 0-2 points;
* Patients with pancreatic ductal adenocarcinoma diagnosed by histology or cytology;
* Expected survival time> 3 months;
* The functions of important organs meet the following requirements;
* The maximum diameter of single lesion ≤ 5cm or the number of multiple lesions ≤ 5 and the maximum diameter ≤ 3cm;
* Measurable lesions that meet RECIST criteria.

  1. Platelet ≥75×109/L, hemoglobin ≥85g/L，white blood cell ≥ 3.0 × 109 / L;
  2. Total bilirubin ≤ 1.5 times upper limit of normal value (ULN) ; ALT and AST ≤ 5 times ULN ;
  3. Albumin ≥ 28g / L;
  4. Creatinine ≤ 1.5 times ULN, or creatinine clearance rate ≥ 50ml / min;
* Women of childbearing age must undergo a negative pregnancy test (βHCG) before starting treatment. Women and men of childbearing age (sexual relationships with women of childbearing age) must agree to use them effectively during treatment and 3 months after the last dose of treatment Contraceptive measures;
* Signature of patient information and informed consent.
* Patients who did not participate in other clinical trials within 4 weeks before screening; those who failed in other trials but met the requirements of this trial could be enrolled.

Exclusion Criteria:

* Patients with distant metastasis include but not limited to lung metastasis, bone metastasis and brain metastasis;
* Other serious diseases or conditions, including congestive heart failure (NYHA grade III or IV), unstable angina, myocardial infarction and cerebral infarction in the past 6 months, severe arrhythmia, prolonged QT interval, active HIV infection or HIV disease, mental disorders, drug abuse, etc;
* Women who are pregnant or nursing, or have fertility but refuse to take contraceptive measures;
* During the enrollment period, a serious active infection requiring antibiotic intravenous treatment occurred;
* In addition to cervical carcinoma in situ, basal cell carcinoma and superficial bladder tumor (TA, tis & T1). Any cancer cured for more than 3 years before enrollment was allowed to be enrolled;
* Patients who cannot follow the trial protocol or cannot cooperate with follow-up;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
OS | 24months
  Overall survival

SECONDARY OUTCOMES:
6-month PFS | 6months
  From date of starting treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
ORR | From the first drug administration up to two years
  Overall Response Rate
DCR | From the first drug administration up to two years
  Disease Control Rate
Complete ablation rate | From the first drug administration up to two years
  The complete ablation rate was evaluated by abdominal enhanced MRI or CT at 4 weeks after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Pelzer U, Opitz B, Deutschinoff G, Stauch M, Reitzig PC, Hahnfeld S, Muller L, Grunewald M, Stieler JM, Sinn M, Denecke T, Bischoff S, Oettle H, Dorken B, Riess H. Efficacy of Prophylactic Low-Molecular Weight Heparin for Ambulatory Patients With Advanced Pancreatic Cancer: Outcomes From the CONKO-004 Trial. J Clin Oncol. 2015 Jun 20;33(18):2028-34. doi: 10.1200/JCO.2014.55.1481. Epub 2015 May 18. PMID 25987694
- [Background] Frampas E, David A, Regenet N, Touchefeu Y, Meyer J, Morla O. Pancreatic carcinoma: Key-points from diagnosis to treatment. Diagn Interv Imaging. 2016 Dec;97(12):1207-1223. doi: 10.1016/j.diii.2016.07.008. Epub 2016 Aug 24. PMID 27567314
- [Background] Kamisawa T, Wood LD, Itoi T, Takaori K. Pancreatic cancer. Lancet. 2016 Jul 2;388(10039):73-85. doi: 10.1016/S0140-6736(16)00141-0. Epub 2016 Jan 30. PMID 26830752
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Tahara J, Shimizu K, Otsuka N, Akao J, Takayama Y, Tokushige K. Gemcitabine plus nab-paclitaxel vs. FOLFIRINOX for patients with advanced pancreatic cancer. Cancer Chemother Pharmacol. 2018 Aug;82(2):245-250. doi: 10.1007/s00280-018-3611-y. Epub 2018 May 30. PMID 29846765
- [Background] Yu X, Gu J, Fu D, Jin C. Dose surgical resection of hepatic metastases bring benefits to pancreatic ductal adenocarcinoma? A systematic review and meta-analysis. Int J Surg. 2017 Dec;48:149-154. doi: 10.1016/j.ijsu.2017.10.066. Epub 2017 Nov 6. PMID 29081375
- [Background] Frigerio I, Regi P, Giardino A, Scopelliti F, Girelli R, Bassi C, Gobbo S, Martini PT, Capelli P, D'Onofrio M, Malleo G, Maggino L, Viviani E, Butturini G. Downstaging in Stage IV Pancreatic Cancer: A New Population Eligible for Surgery? Ann Surg Oncol. 2017 Aug;24(8):2397-2403. doi: 10.1245/s10434-017-5885-4. Epub 2017 May 17. PMID 28516291
- [Background] Hackert T, Niesen W, Hinz U, Tjaden C, Strobel O, Ulrich A, Michalski CW, Buchler MW. Radical surgery of oligometastatic pancreatic cancer. Eur J Surg Oncol. 2017 Feb;43(2):358-363. doi: 10.1016/j.ejso.2016.10.023. Epub 2016 Nov 9. PMID 27856064
- [Background] Park JB, Kim YH, Kim J, Chang HM, Kim TW, Kim SC, Kim PN, Han DJ. Radiofrequency ablation of liver metastasis in patients with locally controlled pancreatic ductal adenocarcinoma. J Vasc Interv Radiol. 2012 May;23(5):635-41. doi: 10.1016/j.jvir.2012.01.080. PMID 22525021
- [Background] Lee SJ, Kim JH, Kim SY, Won HJ, Shin YM, Kim PN. Percutaneous Radiofrequency Ablation for Metachronous Hepatic Metastases after Curative Resection of Pancreatic Adenocarcinoma. Korean J Radiol. 2020 Mar;21(3):316-324. doi: 10.3348/kjr.2019.0647. PMID 32090524